CLINICAL TRIAL: NCT07122700
Title: Non-Invasive Biomarkers for Metabolic Liver Disease (NIMBLE) Study 2.0 - An FNIH Biomarkers Consortium Study
Brief Title: Evaluation of Non-Invasive Tests for Metabolic Liver Disease
Acronym: NIMBLE
Status: Recruiting | Type: Observational
Sponsor: Foundation for the National Institutes of Health (Other)
Responsible Party: Sponsor
Other Study IDs: NIMBLE Study 2.0
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Associated Fatty Liver Disease; Metabolic Associated Steatotic Liver Disease; Cirrhosis, Liver; NASH; Liver Fibrosis; Liver Fat; Liver Steatoses; Liver Inflammation
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected for biomarker analyses, and liver biopsies are obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Non-Invasive Biomarkers for Metabolic Liver Disease (NIMBLE) study is a comprehensive, multi-year collaborative effort to standardize, validate and advance the regulatory qualification of blood- and imaging-based biomarkers to diagnose and stage Metabolic dysfunction-associated steatohepatitis (MASH), previously known as nonalcoholic steatohepatitis (NASH). MASH is characterized by liver inflammation accompanied by simultaneous fat accumulation in the liver.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD), previously known as nonalcoholic fatty liver disease (NAFLD), is a common liver problem which affects 30% of the United States population. Liver biopsy-based histopathology is accepted as the most accurate technique to detect patients at risk of developing serious liver conditions secondary to non-alcoholic steatohepatitis (MASH). However, the liver biopsy is an invasive test with risk for complications and even risk of mortality. Alternative non-invasive blood-based and imaging biomarkers are needed to replace liver biopsy for diagnosis and staging of MASH with fibrosis with the ultimate goal to guide timely decisions for clinical care including pharmacologic intervention for patients with MASH.

The Non-Invasive Biomarkers for Metabolic Liver Disease (NIMBLE) project was commissioned by the FNIH to qualify non-invasive tests (NITs) for MASLD. It represents a collaborative effort involving the FNIH, Food and Drug Administration (FDA), academics and multiple industry partners to qualify biomarkers for diagnosis and staging of MASH with fibrosis. The NIMBLE project plan was designed to occur across two stages (Stage 1 and Stage 2) and with the ultimate goal to generate data on blood-based, Vibration Controlled Transient Elastography- (VCTE) based and imaging-based biomarkers to support seeking regulatory approval of one or more biomarker(s) or biomarker panel(s) for diagnosis and staging of MASH.

Data generated within NIMBLE Stage 1 were able to successfully identify a set of candidate blood-based and imaging biomarkers that met prespecified criteria for further evaluation in Stage 2. The current study aims to deliver on that goal for NIMBLE Stage 2, namely, to confirm and extend the findings from NIMBLE Stage 1 in the setting of a prospective non-interventional trial in a population at risk for MASH with fibrosis. To that end, NIMBLE Study 2.0 is primarily designed to evaluate the performance characteristics of prespecified blood-based, VCTE-based and imaging-based biomarker(s) and biomarker panel(s) when calibrated against liver biopsy-based histology as well as currently available tools for diagnosis and staging of MASH in those at risk.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged > 18 years and < 75 years
4. Participants must exhibit some manifestations of metabolic dysregulation. Either:

A. Physician-diagnosed T2DM for at least 90 days with HbA1c > 6.5 and antidiabetic therapy, if any, stable for at least 90 days prior to screening or B. At least any one of the following six metabolic syndrome criteria [6]

1. body mass index (BMI) of > 25 kg/m2 2. waist circumference: i. > 102 cm for men ii. > 88.9 cm for women 3. fasting triglyceride concentration > 150 mg/dL i. or ongoing treatment with triglyceride lowering medication 4. HDL-cholesterol concentration: i. < 40 mg/dL for men ii. < 50 mg/dL for women iii. or ongoing treatment with cholesterol lowering medication. 5. fasting glucose concentration > 100 mg/dL 6. either semi-recumbent or supine blood pressure systolic > 130 mmHg and/ or diastolic > 85 mmHg i. or ongoing treatment with antihypertensive medication. 5. FIB-4 > 1.3 (age < 65 years) and > 2.0 (age > 65 years) 6. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

1. Known history or evidence of other forms of chronic liver disease other than MASLD/MASH including but not limited to viral hepatitis B or C, autoimmune liver disease, primary biliary cholangitis, primary sclerosing cholangitis, Wilson disease, hemochromatosis, drug-induced liver disease, conditions involving bile duct obstructions, liver cancer, past history of HCC or HCC treatment, listed for or history of liver transplantation, prior resection of liver, etc.
2. Current or past evidence of decompensated liver disease defined by overt ascites that is clinically obvious and requires diuretic therapy, overt encephalopathy requiring therapy or history of variceal hemorrhage
3. Circulating Alanine aminotransferase (ALT)> 5xULN
4. Ongoing or recent (within the last two years prior to screening) consumption of significantly greater than moderate amounts of alcohol.

   * A standard alcoholic drink is any drink that contains about 14 g of pure alcohol, such as 12 fluid ounces of regular beer 8-10 fluid ounces of malt liquor or flavored malt beverages such as hard seltzer 5 fluid ounces of table wine 3-4 fluid ounces of fortified wine such as sherry or port 2-3 fluid ounces of cordial liqueur or aperitif 1.5 fluid ounces (a single jigger or shot) of brandy, cognac, or distilled spirits such as gin, rum, tequila, vodka, whiskey, etc.
   * Significantly greater than moderate alcohol consumption is defined as on average over a 2-year period prior to screening:

   Women
   * >1 standard drink per day and/or
   * >14 standard drinks per week Men
   * >2 standard drinks per day and/or
   * >21 standard drinks per week in men

     * An Alcohol Use Disorders Identification Test (AUDIT) score of 7 or higher
     * A PEth test score of ≥ 20ng/ml.
5. In the opinion of the investigator, any contraindications to liver biopsy including but not limited to having significant uncorrected coagulopathy or thrombocytopenia, on chronic anticoagulation with Direct Oral Anticoagulants (DOACs), or on low dose heparin or Warfarin.
6. Uncontrolled systolic blood pressure > 180 mmHg and diastolic blood pressure > 120 mmHg at screening. Blood pressure will be obtained after at least 10 minutes of resting in a semi-recumbent or supine position.
7. Any systemic disease that in the opinion of the investigator precludes inclusion of the patient in the trial
8. Unable or unwilling to provide informed consent
9. Unwilling to undergo liver biopsy procedure
10. Unable or unwilling to comply with requirements for study procedures (such as fasting)
11. Unable to perform study procedures in the opinion of the investigator
12. Participants who are unwilling or unable (e.g. due active implants such as pacemaker or having a waist diameter (calculated as: diameter = circumference / π) 70cm, unless a wide-bore MRI machine is available) to undergo MRI procedures.
13. Pregnancy or planned pregnancy within 4 months of screening.
14. Participation in another clinical trial within 30 days, or dosing with an investigational agent within 90 days prior to signing the ICF for this study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll participants with suspected or confirmed diagnosis of MASLD.
  Sex: Male and female participants Age: ≥ 18 and < 75 years Population sample: Patients with a high probability of MASLD based on eligibility criteria (details under inclusion/exclusion criteria in Section 5.1) General health status: Patients with suspected or confirmed diagnosis of MASLD and no contraindications precluding participation in any study procedures.
  Geographic location: United States, multi-site
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Detection of At-Risk MASH | within 120 days of study enrollment.
  Evaluate the diagnostic performance of individual and combined biomarkers (e.g., NIS2+, ADAPT [PRO-C3-based score], MRI-AST (MAST) [MRE + PDFF + AST], FAST and Metabolomics-Advanced Steatohepatitis Fibrosis (MASEF) [included in the OWLiver Test]) for identifying at-risk MASH (MASH + MAS ≥4 + fibrosis stage ≥2).
Fibrosis Staging | within 120 days of study enrollment.
  Assess blood-based, imaging, and composite biomarkers (e.g., Enhanced Liver Fibrosis (ELF) Test, Liver Stiffness Measure (LSM) by VCTE, MRE, Agile 3+, Agile 4) for detecting clinically significant fibrosis (≥2), advanced fibrosis (≥3), and fibrosis stage 4 (cirrhosis, histologically defined).
Liver Fat Content Monitoring | within 120 days of study enrollment.
  Evaluate imaging-based biomarkers (e.g., MRI-PDFF, Hepatorenal Index, Controlled Attenuation Parameter (CAP)) for hepatic steatosis monitoring.
Diagnostic Enrichment | within 120 days of study enrollment.
  Identify biomarkers that enhance participant selection for clinical trials, focusing on populations with at-risk MASH, specific fibrosis stages, or steatosis.
Exploratory Biomarkers | within 120 days of study enrollment.
  Investigate exploratory biomarkers (e.g., AI-based histological scoring, sequential testing strategies) for novel diagnostic workflows.

SECONDARY OUTCOMES:
Comparison to Fibrosis (FIB)-4 or other fibrosis-related standards | within 120 days of study enrollment.
  To compare the performance characteristics of one or more 1) blood-based biomarkers, 2) imaging-based biomarkers, 3) VCTE-based biomarkers and 4) multiparametric biomarkers to to FIB-4 or other fibrosis-related standards specific to the context of use (COU) for fibrosis in a population at risk for MASH with fibrosis.
Comparison to ALT or other activity-related standards. | within 120 days of study enrollment.
  To compare the performance characteristics of one or more 1) blood-based biomarkers, 2) imaging-based biomarkers, 3) VCTE-based biomarkers and 4) multiparametric biomarkers to ALT or other activity-related standards specific to the context of use (COU) of at-risk MASH in a population at risk for MASH with fibrosis.
Comparison to Histology. | within 120 days of study enrollment.
  To compare the performance characteristics of one or more 1) blood-based biomarkers, 2) imaging-based biomarkers, 3) VCTE-based biomarkers and 4) multiparametric biomarkers to histology standards to the context of use (COU) for steatosis in a population at risk for MASH with fibrosis.
AI-driven histology endpoints | within 120 days of study enrollment.
  a. Correlation of AI-based digital pathology results with traditional histological scoring systems (MAFLD Activity Score (MAS), fibrosis stages).

CONTACTS AND LOCATIONS:
Overall Officials: Arun Sanyal, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Ohio Clinical Trials, Columbus, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
NIMBLE has an ancillary studies protocol which governs all requests for use of data, beyond the primary publication by project team members who have contributed services to the project. For example, this request covers clinical data that are associated with the biospecimens each company obtained and analyzed, as well as biomarker values, imaging results, and biopsy results generated by project team members.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made publicly available upon closeout (estimated Q4 2026). Until that point, all data are governed by the ancillary studies policy.
Access Criteria: Companies only get access to data they generated and associated clinical values, unless requested via ancillary studies protocol. Project team members who funded the project get access to all IPD.